CLINICAL TRIAL: NCT07052760
Title: Imaging of Solid Tumors Using DLL3 SPECT
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Thomas Hope (Other)
Collaborators: Abdera Therapeutics Inc. (Industry)
Responsible Party: Sponsor-Investigator, Thomas Hope, Professor In Residence, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 25926; NCI-2025-04590 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2025-06-28; First posted 2025-07-07 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Solid Tumor Cancer; Castration Resistant Prostate Cancer; Castration Resistant Prostate Cancer (CRPC); Neuroendocrine (NE) Tumors
Keywords: Imaging Agent Study
MeSH Terms: conditions — Neoplasms | interventions — Immunoconjugates

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cohort 1: Castration resistant prostate cancer (Experimental): Participants will receive a single administration of 185 megabecquerels (MBq) (5 millicurie (mCi)) +/- 10% of 111In-ABD147 prior to SPECT/CT imaging 48 hours after injection. Repeat administration of 111In-ABD147 and SPECT/CT imaging may be performed. Participants will be followed for up to 7 days after the injection of 111In-ABD147 for evaluation of adverse events.
  Interventions: Drug: 111In-ABD147; Procedure: Single-photon emission computed tomography (SPECT)/Computerized tomography (CT)
- Cohort 2: High grade neuroendocrine tumor (Experimental): Participants will receive a single administration of 185 MBq (5 mCi) +/- 10% of 111In-ABD147 prior to SPECT/CT imaging 48 hours after injection. Repeat administration of 111In-ABD147 and SPECT/CT imaging may be performed. Participants will be followed for up to 7 days after the injection of 111In-ABD147 for evaluation of adverse events.
  Interventions: Drug: 111In-ABD147; Procedure: Single-photon emission computed tomography (SPECT)/Computerized tomography (CT)
- Cohort 3: Agnostic solid tumors (Experimental): Participants will receive a single administration of 185 MBq (5 mCi) +/- 10% of 111In-ABD147 prior to SPECT/CT imaging 48 hours after injection. Repeat administration of 111In-ABD147 and SPECT/CT imaging may be performed. Participants will be followed for up to 7 days after the injection of 111In-ABD147 for evaluation of adverse events.
  Interventions: Drug: 111In-ABD147; Procedure: Single-photon emission computed tomography (SPECT)/Computerized tomography (CT)

INTERVENTIONS:
Drug: 111In-ABD147 — Given intravenously (IV) prior to imaging
  Other Names: Radioimmunoconjugate
Procedure: Single-photon emission computed tomography (SPECT)/Computerized tomography (CT) — Undergo imaging
  Other Names: SPECT/CT

SUMMARY:
This is a single arm, pilot trial that evaluates the ability of a novel imaging agent (111In-ABD147) to detect metastatic cancer in participants with solid tumors. 111In-ABD147 is a high affinity Delta-like ligand 3 (DLL3) antigen binding domain fused to an engineered humanized Fc to create an antibody (VHH-Fc) that is bio-conjugated with a DOTA linker-chelator to a 111In radiometal. DLL3 is expressed on a variety of tumors, particularly those with neuroendocrine features.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

1) Determine the feasibility of detecting tumor uptake using 111In-ABD147.

SECONDARY OBJECTIVE:

1) Safety of 111In-ABD147.

EXPLORATORY OBJECTIVES:

1. Correlation of 111In-ABD147 uptake with DLL3 expression determined by immunohistochemistry.
2. Compare 111In-ABD147 scan results to archival Fluorodeoxyglucose (FDG)-Positron Emission Tomography (PET) images when available.

OUTLINE:

Participants will be assigned to cohorts based on solid tumor diagnosis. All participants will receive 1 dose of study drug followed by single-photon emission computed tomography (SPECT)/Computerized tomography (CT) imaging. Repeat administration of 111In-ABD147 and SPECT/CT imaging may be performed. Participants will be followed for up to 7 days after last dose for safety.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Histopathologically confirmed solid tumors in one of the following cohorts:

   1. Cohort 1 (n=15): Histologically confirmed prostate cancer, with castration resistant disease per Prostate Cancer Clinical Trials Working Group 3 (PCWG3) criteria.
   2. Cohort 2 (n=15): Histologically confirmed high grade neuroendocrine tumor, with a Ki-67 over 20.
   3. Cohort 3 (n=15): Agnostic to tumor type.
3. Metastatic disease present on conventional imaging defined as having Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 measurable disease or multiple bone metastases.
4. Ability to understand a written informed consent document, and the willingness to sign it.

Exclusion Criteria:

1. Unlikely to comply with protocol procedures, restrictions and requirements and judged by the Investigator to be unsuitable for participation.
2. Has known hypersensitivity to Chinese hamster ovary cell products.
3. Has a history of severe allergic anaphylactic reactions to chimeric or humanized antibodies or fusion proteins.
4. Known pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-11-30 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Standardized Uptake Values (SUVs) | 2 days
  Standardized Uptake Values (SUVs) will be calculated for up to five lesions in each patient, with mediastinal blood pool being used as background activity. The median and range will be reported across all Response Evaluation Criteria in Solid Tumors (RECIST) measurable lesions broken down by location (organ metastases, nodal metastases and bone metastases).
Tumor-to-background ratio (TBR) | 2 days
  Tumor-to-background ratios (TBR) ratios will be calculated for up to five lesions in each patient, with mediastinal blood pool being used as background activity. The median and range of the measured TBRs will be reported across all RECIST measurable lesions broken down by location (organ metastases, nodal metastases and bone metastases).

SECONDARY OUTCOMES:
Percentage of participants with treatment-emergent adverse events | Up to 7 days
  The percentage of participants with reported treatment-emergent adverse events and the 95% confidence interval following 111In-ABD147 injection will be descriptively reported, using NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas A Hope, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data may be shared with collaborating sponsors during the course of the study
Supporting Information: Study Protocol, SAP, ICF